CLINICAL TRIAL: NCT01315782
Title: Alveolar Dead Space as Predictor of Multi-organ Failure and Mortality in Medical Intensive Care Patients With Sepsis Requiring Mechanical Ventilation
Brief Title: Alveolar Dead Space as Predictor of Organ Failure in Severe Sepsis
Status: Not yet recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Rosa Estrada Y Martin, Associate Professor - IM, Critical Care, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-10-0555
Record Dates: First submitted 2011-03-08; First posted 2011-03-15 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock; Multi-organ Failure
Keywords: Sepsis; Severe sepsis; Septic shock; Alveolar dead space; Multi-organ failure
MeSH Terms: conditions — Sepsis; Shock, Septic; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multi-organ failure: Alveolar dead space on mechanically ventilated patients with severe sepsis or septic shock.

SUMMARY:
This is an observational study to understand the changes in alveolar dead space in medical critically ill patients with severe infection (severe sepsis) requiring mechanical ventilation and the possibility to predict multi-organ failure.

The measurement of alveolar dead space used to require sophisticated equipment and time. New ventilators have microprocessors that allow rapid mathematical calculation with minimal intervention.

DETAILED DESCRIPTION:
The patient will be followed during their ICU stay up to two weeks while on mechanical ventilation.

Patient will be followed daily for the initial 48 hours and then once per week for 2 weeks while mechanically ventilated.

ELIGIBILITY:
Inclusion Criteria:

* Adults with severe sepsis or septic shock on mechanical ventilation
* Enrolled in the initial six hours of ICU admission

Exclusion Criteria:

* Patients with withdrawal or hospice order.
* Patients with terminal, irreversible disease, expect to decease in 48 hours from ICU admission.
* Patients with COPD.
* Patients transferred from outside ICU with ongoing sepsis management for more than six hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to medical intensive care unit with severe sepsis or septic shock requiring mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Multi-organ failure | daily for 48 hours then weekly for 2 weeks.
  Multi-oran failure will be accessed by daily laboratory data, heart function by echocardiogram if available, urinary output, vitals and use of vasopressors.

SECONDARY OUTCOMES:
Mortality | ICU mortality
  All the patient will be followed up to 28-days to determine survival.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Estrada-Y-Martin, MD MSc, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States